CLINICAL TRIAL: NCT00387686
Title: A Phase 2/3, Multicenter, Double-Blind, Randomized, Controlled Study Of Recombinant Human Bone Morphogenetic Protein-2 (rhBMP-2)/Calcium Phosphate Matrix (CPM) In Closed Diaphyseal Tibial Fracture
Brief Title: A Phase 2/3 Multicenter, Controlled Trial Of rhBMP-2/CPM In Tibial Fractures
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decision was taken by Wyeth Sr. Management to early terminate the 3100N7-210 study (terminate enrollment but complete follow-up).
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3100N7-210
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Fractures
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): 1.0 mg/mL rhBMP-2/CPM + surgical fixation
  Interventions: Drug: rhBMP-2/CPM
- B (Experimental): 2.0 mg/mL rhBMP-2/CPM + surgical fixation
  Interventions: Drug: rhBMP-2/CPM
- C (Active Comparator): Buffer/CPM + surgical fixation Intervention
  Interventions: Drug: rhBMP-2/CPM
- D (Other): Standard of Care: Surgical fixation intervention
  Interventions: Drug: rhBMP-2/CPM

INTERVENTIONS:
Drug: rhBMP-2/CPM
  Arms: A
Drug: rhBMP-2/CPM
  Arms: B
Drug: rhBMP-2/CPM
  Arms: C
Drug: rhBMP-2/CPM
  Arms: D

SUMMARY:
The primary objective of this study is to assess whether a single dose of rhBMP-2/CPM administered at the fracture site via percutaneous injection, in combination with standard of care, accelerates fracture union and return to normal function in subjects who have a closed diaphyseal tibial fracture when compared to standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature, male and female subjects who are at least 18 years old.
* Closed diaphyseal tibial fracture.
* Closed reduction and definitive internal fixation by means of a reamed, locked intramedullary nail within 72 hours after injury.

Exclusion Criteria:

* Concurrent fractures of the ipsilateral or contralateral lower extremity other than the ipsilateral fibula, that would impede performance on the functional assessment of weight bearing.
* Planned procedure(s) to stimulate fracture healing after intramedullary nailing.
* Neurovascular impairment of the fractured limb, deep vein thrombosis, or (impending) compartment syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess whether a single dose of rhBMP-2/CPM administered in combination with the SOC accelerates fracture union and return to normal function as indicated on radiographs and functional evaluations. | efficacy will be demonstrated if there is a greater than or equal to 4 week reduction in time to fra

SECONDARY OUTCOMES:
Demonstrate safety of rhBMP-2/CPM administration; demonstrate earlier return to function; assess feasibility of rhBMP-2CPM administration. Subject enrollment 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (16):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Portage, Michigan
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Elmhurst, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
- Pfizer Investigational Site, Buenos Aires, Argentina
- Australia (4):
  - Pfizer Investigational Site, Liverpool, New South Wales
  - Pfizer Investigational Site, New Lambton, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
- Brazil (2):
  - Pfizer Investigational Site, Cerequeira Cesar, São Paulo
  - Pfizer Investigational Site, Vila Clemetino, São Paulo
- Canada (6):
  - Pfizer Investigational Site, Ajax, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Scarborough Village, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Finland (2):
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Turku
- France (4):
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Toulouse
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Münster
- India (5):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
- Pfizer Investigational Site, Riga, Latvia
- Mexico (5):
  - Pfizer Investigational Site, Chihuahua City, Chihuahua
  - Pfizer Investigational Site, Col. Los Morales, Del Miguel, Hidalgo
  - Pfizer Investigational Site, Col. El Retiro, Guadalajara, Jal.
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Guadalajara, Jal
- Poland (2):
  - Pfizer Investigational Site, Bielsk Podlaski
  - Pfizer Investigational Site, Krakow
- Romania (3):
  - Pfizer Investigational Site, Cluj-Napoca, Cluj
  - Pfizer Investigational Site, Iași, Iaşi
  - Pfizer Investigational Site, Bucharest
- Serbia (2):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Niš
- Pfizer Investigational Site, Ljubljana, Slovenia
- Spain (3):
  - Pfizer Investigational Site, Alcalá de Henares, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Alcalá
- Pfizer Investigational Site, Uppsala, Sweden
- United Kingdom (2):
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Norwich

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3100N7-210&StudyName=A%20Phase%202/3%20Multicenter%2C%20Controlled%20Trial%20Of%20rhBMP-2/CPM%20In%20Tibial%20Fractures